CLINICAL TRIAL: NCT05047380
Title: The Relationship of Disability With Depression, Anxiety and Sleep Quality in Patients With Coccygodynia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Emel Güler, Associate Professor, Cumhuriyet University
Other Study IDs: 2021-06/20
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Coccyx Injuries; Pain, Chronic; Anxiety; Depression; Sleep; Sleep Hygiene
Keywords: coccyx; chronic pain; depression; anxiety; sleep hygiene
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Depression; Sleep Hygiene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- coccycodinia group: A total of 54 patients diagnosed with coccycodinia
  Interventions: Behavioral: Owstery Disability Scale for disability Beck Depression Scale, Beck Anxiety Scale for psychological evaluation, VAS for pain, Pittsburgh Sleep Quality Scale for sleep quality

INTERVENTIONS:
Behavioral: Owstery Disability Scale for disability Beck Depression Scale, Beck Anxiety Scale for psychological evaluation, VAS for pain, Pittsburgh Sleep Quality Scale for sleep quality — All assessments will be made using questionairres. The Oswestry Disability Index scale will be filled in to assess the severity of disability resulting from pain in the patient. Pain severity will be evaluated with the Visual Analog Scale (VAS). Depression and anxiety assessment will be made with Beck Depression Scale and Beck Anxiety Scale, respectively. Sleep quality will be evaluated with the Pittsburg Sleep Quality Index.

SUMMARY:
Pain of the sacrococcygeal region is called coccygodynia This painful clinical picture, which causes a decrease in the quality of life, also causes disability. Coccycodynia has been associated with hysteria, neurosis, and depression. In some studies, it has been reported that it should be evaluated in somatization in coccygodynia. There are a few studies examining the relationship between coccygodynia and psychiatric disorders.There is no study in the literature examining coccygodynia and sleep. There may be a relationship between pelvic floor muscle spasm in the etiology of coccygodynia and sleep quality. In this study, it is aimed to investigate the relationship between disability severity and anxiety, depression and sleep quality in patients with coccygodynia.

DETAILED DESCRIPTION:
Coccygodynia often develops from an inappropriate sitting position or when standing up from a sitting position. In the advanced stages of coccygodynia the pain becomes continuous. Pain can be triggered by walking or standing for a long time. Patients may experience sacrococcygeal pain in the supine position and during sleep. It has been argued that the coexistence of coccygodynia and psychiatric disease is caused by the excessive activity of the pelvic region nerves. In addition, it has been stated that stress, depression and fear may lead to increased spasm in the pelvic floor muscles.It is stated in the literature that 62.9-75% of patients with chronic pain have at least one psychiatric disorder. The most common psychiatric comorbidities in patients with chronic pain are; major depression, somatoform disorders, and generalized anxiety disorder. The relationship between pain and psychological variables has been attributed to the fact that the sensorial pathways of pain and mood regulation are located in the same region of the brain. In addition, common neurotransmitters such as serotonin, norepinephrine and dopamine are present in the pathophysiology of depression and pain.There is a bidirectional relationship between sleep and pain. In recent studies; It has been reported that sleep disorder causes pain development rather than the effect of pain on sleep disorder.

54 patients with coccydynia will be recruited prospectively according to the appropriate inclusion and exclusion criteria.Within the scope of the study, the age, gender, duration of symptoms, etiology of coccygodynia, and severity of pain will be recorded. The Oswestry Disability Index scale will be filled in to assess the severity of disability resulting from pain in the patient. Pain severity will be evaluated with the Visual Analog Scale (VAS). Depression and anxiety assessment will be made with Beck Depression Scale and Beck Anxiety Scale, respectively. Sleep quality will be evaluated with the Pittsburg Sleep Quality Index.

The data will be entered into the SPSS (version: 22.0) IBM SPSS statistical package program. Arithmetic mean, standard deviation, min-max, median values will be given in the data obtained by measurement. Percentage and frequency distribution will be given in the data obtained by counting. In statistical evaluations, parametric tests will be used for normally distributed data, and non-parametric tests will be used for data not normally distributed. Relationships will be compared according to the Pearson or Spearman correlation coefficient. Chi-square test will be applied to categorical data. P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coccygodynia
* Agreement to take part in the study 18 to 70 years old

Exclusion Criteria:

* Presence of cognitive impairment that would limit answering the questions in the questionnaires
* History of psychotic disorder
* History of neurological disease (cerebrovascular accident, polyneuropathy, parkinson's, dementia, epilepsy),
* History of rheumatological disease, fibromyalgia and malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Sivas Cumhuriyet University Faculty of Medicine, Physical Therapy and Rehabilitation Clinic between 01/08/2021-30/04/2022 and diagnosed with coccygodynia will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression | The study will be completed in 9 months.
  Beck Depression Scale will be used in depression interrogation. ≤9 points are classified as normal,10-16 points as mild depression,17-29 points as moderate depression, and 30-63 points as severe depression.Beck Anxiety Scale will be used in anxiety interrogation. ≤9 points are classified as normal, 10-18 points as mild anxiety, 19-29 points as moderate anxiety, and 30-63 points as severe anxiety.
Sleep quality | The study will be completed in 9 months.
  Sleep quality will be questioned with The Pittsburgh Sleep Quality Index. Those who score ˃5 have poor sleep quality, and those who score ≤5 have "good sleep quality".

CONTACTS AND LOCATIONS:
Overall Officials: Emel Güler, MD, Principal Investigator — Cumhuriyet University
Locations (1):
- Emel Guler, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanley EN, Ode G, Jackson Iii BJ, Seymour R. Coccygectomy for patients with chronic coccydynia: a prospective, observational study of 98 patients. Bone Joint J. 2016 Apr;98-B(4):526-33. doi: 10.1302/0301-620X.98B4.36641. PMID 27037436
- See also: preoperative psychiatric disorders were detected in most of the patients who underwent coccygectomy. — https://pubmed.ncbi.nlm.nih.gov/27037436/